CLINICAL TRIAL: NCT03935022
Title: Anthocyanin Bioavailability and Plasma Antioxidant Capacity in Healthy Volunteers After Acute Rice Intake
Brief Title: Rice Anthocyanin Bioavailability in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Marcello Iriti, Professor, University of Milan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Unimi_DiSAA_01
Record Dates: First submitted 2019-04-17; First posted 2019-05-02 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Black rice Venere (Experimental): Healthy volunteers will receive the black rice Venere in a cross-over randomized clinical trial (after 7 days wash-out).
  Interventions: Other: Rice
- Black rice Artemide (Experimental): Healthy volunteers will receive the black rice Artemide in a cross-over randomized clinical trial (after 7 days wash-out).
  Interventions: Other: Rice
- Complete white rice (Sham Comparator): Healthy volunteers will receive the complete white rice in a cross-over randomized clinical trial (after 7 days wash-out).
  Interventions: Other: Rice

INTERVENTIONS:
Other: Rice — Each group will randomly receive, during three different experimental days, one of the following treatments by different allocation sequences:
  1. 80g of black rice Venere (Group A)
  2. 80g of black rice Artemide (Group B)
  3. 80g of brown rice (Group C) The three treatments will be separated by a 7 day wash-out period. After an overnight fast, volunteers will consume the rice serving within 10-15 min, immediately after the first basal blood collection at 8:00 a.m. (baseline). Other blood withdrawals will be carried out a 0.5, 1.0, 2.0 and 3.0 h after rice administration.

SUMMARY:
Aims of the project

1. To determine the rice anthocyanin content via high-performance liquid chromatographycoupled to mass spectrometry, HPLC-MS
2. To study the oral bioavailability of anthocyanins in healthy volunteers after the intake of a serving (80 g) of black rice (Venere and Artemide varieties).
3. To determine the plasma biokinetics parameters of rice anthocyanins via spectrophometric determination and high-performance liquid chromatographycoupled to mass spectrometry, HPLC-MS.

DETAILED DESCRIPTION:
To limit the interindividual variability, The protocol will be designed as a prospective, randomized, cross-over pharmacokinetic study on healthy volunteers. Participants will be randomly divided into three groups (black rice Venere, black rice Artemide and white rice/control) by an allocation software ( http://graphpad.com/quickcalcs/randomise1.cfm ) which will generate different random sequences of the treatment assignment.

Subjects will be deprived of anthocyanin-rich food sources 7 days before experimentation (wash-out period). Each volunteer will receive a complete list of anthocyanin-rich foods to be avoided, including berry fruits (i.e. blueberries, cranberries, raspberries, blackcurrants and elderberries), red/violet fruits/vegetables (i.e. grapes, cherries, pomegranates, red apples, plums, eggplants, tomatoes and peppers), red wine and other colored products (i.e. marmalade, jams and juices containing berries). Breakfast, lunch and dinner will be standardized 1 day before the experiment. Each group will randomly receive, during three different experimental days, one of the following treatments by different allocation sequences:

1. 80g of black rice Venere (Group A)
2. 80g of black rice Artemide (Group B)
3. 80g of white rice (Group C)

Therefore, each subject will be involved in three experimental days. The three treatments will be separated by a 7 day wash-out period.

After an overnight fast, volunteers will consume the rice serving within 10-15 min, immediately after the first basal blood collection at 8:00 a.m. (baseline). Other blood withdrawals will be collected after 30 minutes, 1 hour, 2 hours, 3 hours.

Chemical analyses. The extraction protocols of anthocyanins from body fluids will be developed, in order to reach the maximum yield of the analytes from the samples. Plasma anthocyanins will be measured by spectrophometric determination and high-performance liquid chromatographycoupled to mass spectrometry, HPLC-MS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy status
* Age: 18-45
* Normal weight (BMI 18.5-24.9) who voluntarily accept to join the study, after informed consent.

Exclusion Criteria:

* <18 Years;
* Pregnancy and lactation;
* Systemic disorders;
* Dietary supplements intake (vitamins, antioxidants, botanicals, phytochemicals)
* Abnormal hematological parameters;
* Heavy smoking and alcohol drinking;
* High-intensity physical activity.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-07-21 (Actual)

PRIMARY OUTCOMES:
Changes in plasma total anthocyanin detection | 0.0 (baseline, before starting the intervention), then after 0.5 hour, 1 hour, 2 hours and 3 hours
  Total anthocyanins will be detected via spectrophometric determination; expressed as μg of catechin per mL of plasma
Changes in plasma Cyanidin-3-O-glucoside detection | 0.0 (baseline, before starting the intervention), then after 0.5 hour, 1 hour, 2 hours and 3 hours
  Cyanidin-3-O-glucoside will be detected via high-performance liquid chromatographycoupled to mass spectrometry, HPLC-MS) in plasma; expressed nM (nano molar) in plasma

SECONDARY OUTCOMES:
Changes in plasma antioxidant capacity ABTS | 0.0 (baseline, before starting the intervention), then after 0.5 hour, 1 hour, 2 hours and 3 hours
  2,2'-azino-bis(3-ethylbenzothiazoline-6-sulfonic acid) (ABTS+); the results are expressed as Trolox equivalent antioxidant capacity (TEAC, mmoleq Trolox/mL plasma)
Changes in plasma antioxidant capacity DPPH | 0.0 (baseline, before starting the intervention), then after 0.5 hour, 1 hour, 2 hours and 3 hours
  2,2-diphenyl-1-picrylhydrazyl (DPPH); percentage of inhibition (I%) is calculated as [(ABScontrol 517 nm - ABSsample 517 nm/ABScontrol 517 nm)×100]

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Iriti, Principal Investigator — University of Milan
Locations (1):
- Marcello Iriti, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Conesa MT, Chambers K, Combet E, Pinto P, Garcia-Aloy M, Andres-Lacueva C, de Pascual-Teresa S, Mena P, Konic Ristic A, Hollands WJ, Kroon PA, Rodriguez-Mateos A, Istas G, Kontogiorgis CA, Rai DK, Gibney ER, Morand C, Espin JC, Gonzalez-Sarrias A. Meta-Analysis of the Effects of Foods and Derived Products Containing Ellagitannins and Anthocyanins on Cardiometabolic Biomarkers: Analysis of Factors Influencing Variability of the Individual Responses. Int J Mol Sci. 2018 Feb 28;19(3):694. doi: 10.3390/ijms19030694. PMID 29495642
- [Background] Krga I, Milenkovic D. Anthocyanins: From Sources and Bioavailability to Cardiovascular-Health Benefits and Molecular Mechanisms of Action. J Agric Food Chem. 2019 Feb 20;67(7):1771-1783. doi: 10.1021/acs.jafc.8b06737. Epub 2019 Feb 8. PMID 30698008
- [Background] Ciulu M, Cadiz-Gurrea ML, Segura-Carretero A. Extraction and Analysis of Phenolic Compounds in Rice: A Review. Molecules. 2018 Nov 6;23(11):2890. doi: 10.3390/molecules23112890. PMID 30404149
- [Background] Dias ALS, Pachikian B, Larondelle Y, Quetin-Leclercq J. Recent advances on bioactivities of black rice. Curr Opin Clin Nutr Metab Care. 2017 Nov;20(6):470-476. doi: 10.1097/MCO.0000000000000417. PMID 28858891
- [Background] Van Hung P. Phenolic Compounds of Cereals and Their Antioxidant Capacity. Crit Rev Food Sci Nutr. 2016;56(1):25-35. doi: 10.1080/10408398.2012.708909. PMID 25075608